CLINICAL TRIAL: NCT05742152
Title: Between-day Reliability and Concurrent Validity of Outcome Measures for Pain in Multiple Sclerosis
Brief Title: Reliability and Validity of Outcome Measures for Pain in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Peter Feys, Prof. dr., Hasselt University
Other Study IDs: B1152022000014
Record Dates: First submitted 2023-01-28; First posted 2023-02-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: Pain, outcome measure, assessment, multiple sclerosis, reliability, validity
MeSH Terms: conditions — Pain; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to provide values of test-retest reliability and insights from concurrent validity of outcome measures for pain in multiple sclerosis.

DETAILED DESCRIPTION:
Pain is one of the most annoying symptoms in multiple sclerosis (MS). However, it is underestimated albeit its high prevalence rate with 63%. It negatively affects health related quality of life, activity of daily living, mental health, social functioning, employment, sleep and life enjoyment. In literature, the prevalence of pain varies in the MS literature from 29% to 86%. This wide-range prevalence is the result of methodological differences and non-uniformity of the studied populations which makes pain unclear and underdiagnosed in multiple sclerosis.It is hypothesized that the consistency, severity and interference of pain have varying relationships between other factors such as depression, anxiety, sleep or fatigue.

Evaluating pain was done with various outcome measures resulting in inconclusive results. However, very few of the pain outcome measures are validated for MS population. Thus, it cannot be advised yet whether they contain similar or complementary information. Finally, the interference of pain on activities and participation level of the International Classification of Functioning, Disability and Health (ICF) is poorly documented.

This project aims to put the foundations for future interventional research by providing values of test-retest reliability and insights from concurrent validity. As well, the perceived interference from pain on activities and participation level will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above,
* Ambulatory pwMS with definite diagnosis based on McDonald criteria
* Expanded Disability Status Scale of 6.0 or below,
* Having pain in last month
* Able to understand and answer the questions in the questionnaires.

Exclusion Criteria:

* Diagnosed with major musculoskeletal disorder and any neurological disorder other than MS,
* a relapse in the last month before enrolment,
* cognitive decline that renders the patient incapable of performing tests and questionnaires,
* patients with only headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with MS with pain
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Douleur Neuropathique 4 (DN4) Questionnaire | Day 1 and day 7
  screening tool

SECONDARY OUTCOMES:
PainDETECT Questionnaire | Day 1 and day 7
  screening tool

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (3):
  - National MS center, Melsbroek, Brabant
  - Noorderhart, Overpelt, Limburg
  - AZ Sint-Jan, Bruges
- Pontificia universidad catolica de Chile, Santiago, Chile

REFERENCES:
- [Derived] Yilmazer C, D'haeseleer M, Soler B, Van Wijmeersch B, Solaro C, Ciampi E, Carcamo C, Van Asch P, Cambron M, Lamers I, Feys P. Assessing pain in multiple sclerosis: Test-retest reliability of patient-reported outcome measures and accuracy of screening tools. Mult Scler. 2025 Apr;31(4):474-488. doi: 10.1177/13524585241310139. Epub 2025 Jan 16. PMID 39819131